CLINICAL TRIAL: NCT05477758
Title: The Impact of Pain on Depression Outcomes of Older Adults in Behavioural Activation: An Exploratory Secondary Data Analysis
Brief Title: The Impact of Pain on Depression Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Teesside University (Other)
Collaborators: University of York (Other)
Responsible Party: Principal Investigator, Alexandra Carne, Chief Investigator, Teesside University
Other Study IDs: 8838; ISRCTN02202951 (Registry Identifier: ISRCTN registry); ISRCTN45842879 (Registry Identifier: ISRCTN registry); ISRCTN95270332 (Registry Identifier: ISRCTN registry)
Record Dates: First submitted 2022-07-12; First posted 2022-07-28 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pain; Depression
Keywords: Older Adults; Behavioural Activation
MeSH Terms: conditions — Pain; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CASPER: A multi-centred, pragmatic, two-arm parallel open RCT. Participants with Subthreshold depression were individually randomised (1:1) to receive either collaborative care focusing on behavioural activation or usual GP care
  Interventions: Behavioral: Collaborative care; Other: Usual General Practitioner (GP) care
- CASPER+: A multi-centred, pragmatic, two-arm parallel open RCT. Participants with Major depression were individually randomised (1:1) to receive either collaborative care focusing on behavioural activation or usual GP care
  Interventions: Behavioral: Collaborative care; Other: Usual General Practitioner (GP) care
- SHARD: A multi-centred, pragmatic, two-arm parallel open RCT. Participants with Subthreshold depression were individually randomised (1:1) to receive the self-help booklet based on the principles of behavioural activation or usual GP care
  Interventions: Other: Usual General Practitioner (GP) care; Behavioral: Behavioral Activation Self-Help guide

INTERVENTIONS:
Behavioral: Collaborative care — Participants in the intervention group were allocated a receive a low-intensity programme of behavioural activation specifically designed for adults ≥65 with subthreshold depression. An allocated case manager (primary care mental health worker/ Improving Access to Psychological Therapy) delivered collaborative care for an intended 8-10 weeks. This ran alongside general practitioner (GP) usual care. Collaborative care in both CASPER and CASPER+ trial included weakly telephone/ face-to-face support, active surveillance and symptom monitoring
  Other Names: behavioural activation
  Groups: CASPER; CASPER+
Other: Usual General Practitioner (GP) care — Participants allocated to the control group received usual GP care. Participants did not receive any additional care to their usual primary care management for subthreshold (CASPER) or Major (CASPER+) depression in line with National Institute for Health and Care Excellence (NICE) guidelines as implemented in their GP and local service provision.
Behavioral: Behavioral Activation Self-Help guide — Participants in the intervention arm were provided with a self-help booklet based on clear principles of BA for depression. The purpose of the booklet was to introduce simple behavioural strategies for improving mood. Participants were encouraged to (1) re-establish their daily routine, (2) increase meaningful activities and (3) reduce avoidance behaviours. Participants also received 3 phone calls at week 1, 3 and 6 designed to check the booklet had arrived and to encourage the use of the materials. All participants received their usual GP care
  Groups: SHARD

SUMMARY:
This study is a secondary data analysis of three of largest Randomised Controlled Trials (RCTs) of behavioural activation (BA) for older people with depression in the United Kingdom (UK) primary care. The analysis will aim to explore the impact of pain on depression outcomes of older people receiving BA and potentially identify sub-groups of people who may not respond as well to treatment.

DETAILED DESCRIPTION:
Previous findings have indicated that pain might be an important barrier in depression treatment both with antidepressant medication and in a United States (US) collaborative care model using problem solving therapy and antidepressant medication. It is unknown, however, if pain impacts depression outcomes of older adults in a collaborative care (CC) framework focusing on a brief psychological intervention of BA. Collectively CASPER, CASPER PLUS (+) and SHARD are three of the largest pragmatic, multi-centre randomised controlled trials (RCT) of BA for older adults in UK primary care with low mood and depression. The purpose of this secondary data analysis is, therefore, to explore if pain moderates (modifies) the effect of BA on depression outcomes in older adults, potentially identifying subgroups of older adults who may not respond as well to BA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in CASPER, CASPER + or SHARD study

Exclusion Criteria:

* Anyone who did not consent into one of the three studies above

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were aged 65 years or older with subthreshold depression (CASPER and SHARD) or case-level depression (CASPER+)
Sampling Method: Non-Probability Sample
Enrollment: 1522 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
PhQ-9 (Patient Health Questionnaire- 9 | Baseline
  5 point likert scale ranging from 0 to 27. Higher points denote worse depression. The instrument is used for screening, diagnosing, monitoring and measuring the severity of depression in primary care.
PhQ-9 (Patient Health Questionnaire- 9 | 4 months
  5 point likert scale ranging from 0 to 27. Higher points denote worse depression. The instrument is used for screening, diagnosing, monitoring and measuring the severity of depression in primary care.
SF-12 (Short Form- 12) | Baseline
  The instrument is a generic health status measure consisting of 12 questions measuring 8 domains. Question 8 referring to bodily pain will be used for the moderation analysis. The tool has a likhert scale of 1-5 with 5 denotating worse pain.
EQ-5D (Euroqual Group) | Baseline
  The EQ-5D consists of 5 questions assessing the various quality of life dimensions including mobility, self-care, usual activities, Pain/Discomfort and Anxiety/Depression. Each dimension is rated on three levels: no problem (score=1) some problems (score=2) and extreme problems (score=3). Question 4 relating to pain/discomfort will be used as a second indicator for the pain moderator.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra S Carne, PhD Student, Principal Investigator — Teesside University/ Univeristy of York
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bosanquet K, Adamson J, Atherton K, Bailey D, Baxter C, Beresford-Dent J, Birtwistle J, Chew-Graham C, Clare E, Delgadillo J, Ekers D, Foster D, Gabe R, Gascoyne S, Haley L, Hamilton J, Hargate R, Hewitt C, Holmes J, Keding A, Lewis H, McMillan D, Meer S, Mitchell N, Nutbrown S, Overend K, Parrott S, Pervin J, Richards DA, Spilsbury K, Torgerson D, Traviss-Turner G, Trepel D, Woodhouse R, Gilbody S. CollAborative care for Screen-Positive EldeRs with major depression (CASPER plus): a multicentred randomised controlled trial of clinical effectiveness and cost-effectiveness. Health Technol Assess. 2017 Nov;21(67):1-252. doi: 10.3310/hta21670. PMID 29171379
- [Result] Gilbody S, Brabyn S, Mitchell A, Ekers D, McMillan D, Bailey D, Hems D, Chew Graham CA, Keding A, Bosanquet K; SHARD collaborative. Can We Prevent Depression in At-Risk Older Adults Using Self-Help? The UK SHARD Trial of Behavioral Activation. Am J Geriatr Psychiatry. 2022 Feb;30(2):197-207. doi: 10.1016/j.jagp.2021.06.006. Epub 2021 Jun 19. PMID 34266750
- [Result] Lewis H, Adamson J, Atherton K, Bailey D, Birtwistle J, Bosanquet K, Clare E, Delgadillo J, Ekers D, Foster D, Gabe R, Gascoyne S, Haley L, Hargate R, Hewitt C, Holmes J, Keding A, Lilley-Kelly A, Maya J, McMillan D, Meer S, Meredith J, Mitchell N, Nutbrown S, Overend K, Pasterfield M, Richards D, Spilsbury K, Torgerson D, Traviss-Turner G, Trepel D, Woodhouse R, Ziegler F, Gilbody S. CollAborative care and active surveillance for Screen-Positive EldeRs with subthreshold depression (CASPER): a multicentred randomised controlled trial of clinical effectiveness and cost-effectiveness. Health Technol Assess. 2017 Feb;21(8):1-196. doi: 10.3310/hta21080. PMID 28248154

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT05477758/SAP_001.pdf